CLINICAL TRIAL: NCT03012113
Title: The Effect of Mirabegron on Brown Adipose Tissue in Healthy Young White Caucasian and South Asian Men
Brief Title: Mirabegron and Brown Adipose Tissue
Acronym: Mirab
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ingrid Jazet (Other)
Responsible Party: Sponsor-Investigator, Ingrid Jazet, Dr, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P16.023
Record Dates: First submitted 2016-12-15; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Obesity
Keywords: Adipose tissue; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Short term mild cooling (Other): Subjects will undergo a short term mild cooling protocol consisting of personalized water cooling method for approximately 2 hours.
  Interventions: Other: Short term mild cooling
- Mirabegron (Active Comparator): Subjects will receive one dosage of 200 mg Mirabegron (Astellas Pharma).
  Interventions: Drug: Mirabegron
- Placebo (Placebo Comparator): Subjects will receive one dosage of Placebo, which is packed and labeled to mach the active compound.
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Mirabegron
  Other Names: Betmiga
  Arms: Mirabegron
Other: Short term mild cooling
  Arms: Short term mild cooling
Drug: Placebo Oral Capsule
  Arms: Placebo

SUMMARY:
Obesity and type 2 diabetes (T2D) are emerging problems worldwide. In particular South Asian individuals (representing 20% of the world population) have an increased risk of obesity and related disorders. They are at higher risk for the development of T2D as compared to white Caucasians and develop T2D at a younger age and with lower BMI. The underlying mechanisms that might explain these ethnical differences have not been clarified or understood yet. As a consequence, treatment options are limited and unfocussed, and novel specific strategies are needed.

Brown adipose tissue (BAT) has recently been discovered as a major player in energy metabolism in humans. In a process known as thermogenesis, BAT takes up fatty acids (FA) and glucose from the circulation and subsequently combusts FA and glucose into heat, thereby increasing energy expenditure and improving glucose and FA metabolism. Using 18F-fluorodeoxyglucose (18F-FDG) (positron emission tomography/computed tomography) PET-CT scan analysis investigators have recently shown that South Asian individuals have less brown adipose tissue (BAT) than white Caucasians. This might suggest that they have a lower energy metabolism, which could underlie their increased predisposition for obesity and the development of T2D.

Activation of BAT, for example by cold exposure, was shown to have beneficial metabolic effects in humans. Cold acclimatization can increase BAT volume, nonshivering thermogenesis, glucose uptake by BAT, as well as decrease fat mass in healthy young men. Therefore activation of BAT is considered as a novel therapeutic target in the treatment of obesity and T2D. As cold exposure is not the most desired therapeutic strategy for humans, current pre-clinical research focuses on pharmacological activation of BAT.

β3-receptor agonists can be used to mimic sympathetic innervation of BAT. Our recent studies using mice with a human-like lipoprotein profile showed that treatment with a β3-receptor agonist decreased fat mass, improved dyslipidemia, increased insulin sensitivity and even attenuated the development of atherosclerosis. Likewise, the novel β3-receptor agonist (Mirabegron) has recently been shown to activate BAT in healthy young men as effectively as cold exposure. Therefore, ß3-receptor agonism would be a promising treatment option to activate BAT and enhance energy expenditure, especially for South Asians.

Currently the most common way to visualize BAT in humans is by 18F-FDG PET-CT scan. However this method is both expensive and invasive, as it uses ionizing radiation. Recently, MRI, which has no radiation burden, has emerged as a novel method to visualize BAT in humans. Activation of BAT results in combustion of intracellular lipid stores, which eventually leads to a lower triglyceride (TG) content. MRI can measure TG content of tissue, and using MRI technology the activation of BAT can be quantified by the relative reduction in the TG content of BAT. The use of MRI to visualize and quantify BAT activity is a safe, cost-effective and innovative alternative to PET-CT, which has a potential to become a new gold standard in the nearby future.

To investigate whether β3-receptor agonism has therapeutic potential to improve the metabolic phenotype of South Asians, investigators will perform a randomized cross-over study in which 20 healthy young men aged 18-30 years with a lean body type (BMI <25 kg/m2) are included. Dutch South Asian individuals (n=10) and matched Dutch white Caucasian individuals (n=10) will participate in a cross-over study consisting of three different regimes.

This study will investigate whether β3-receptor agonism has therapeutic potential to improve the metabolic phenotype of South Asians. The effects of a β3-receptor agonist on BAT activity in South Asians have never been studied before. Elucidating the effects of this β3-receptor agonist on BAT activity in South Asians might have major clinical implications, as it might result in the discovery of a potential novel treatment strategy to combat obesity and T2D in this especially vulnerable population.

DETAILED DESCRIPTION:
In the current study, the effect of one single dose of Mirabegron (200 mg) versus placebo and cold-exposure will be studied in health young (18-30 years) Dutch South Asian (n=10) and Dutch Caucasian (n=10) men.

All study subjects will be screened. If the subject meets all the inclusion criteria, is willing to participate in the study and has signed the informed consent, he will be included. All subjects will be asked not to make any changes in their usual diets and physical activities before the start of the whole study.

At screening a thorough medical history and physical examination will be performed. Subjects will be examined while in the fasting state. Anthropometric measurements will be performed as well as a BIA measurement for determination of body fat percentage and basal blood sample will be taken by means of a venapunction. Basal blood measurements include kidney, liver, thyroid, hemoglobulin, natrium, kalium, ureum and lipid parameters as well as glucose concentrations.

If subjects are eligible to participate they first will complete Study day 1, on which we will measure BAT activity and volume before and after cold exposure. Subject will undergo a baseline oxycon and finapres measurement to determine REE and blood pressure and heart rate (30 min). After this a baseline MRI scan will be made followed by an individualized cooling protocol so that the maximum non-shivering thermogenesis is reached. During the cold exposure, skin temperature will be measured via 'iButtons'. One iButtons will be placed under the armpit as an approximation of the 'core temperature'. When shivering temperature is reached, stable cooling period will start (t=0). After 30 minutes of stable cold exposure (t=30) REE and blood pressure and heart rate will be analyzed a second time using a ventilated hood system and the finapres. Thereafter (t=60) BAT activity and volume will be measured using a second MRI scan. Furthermore, during the cooling procedure a venous blood sample will be obtained every 15 minutes to monitor dynamic changes in plasma lipids. In addition, plasma catecholamine concentrations will be determined. If there is no increased BAT activity upon cold stimulation the subject will be excluded from further participation in the study. If there is detectable BAT activity on Study day 1, subjects will participate in Study days 2 and 3 and will be randomized to receive first Mirabegron or placebo to minimize bias.

On study day 2 first baseline oxycon and finapres measurements will be performed to determine REE and blood pressure and heart rate (30 min). Thereafter, the subject will receive a single dose of 200 mg Mirabegron (four tables of 50 mg) (or placebo) (t=0). Again skin temperature will be measured via 'iButtons'. One iButton will be placed under the armpit as an approximation of the 'core temperature'. After 1, 2 and 3 hours (t=60, t=120 and t=180) REE is analyzed using a ventilated hood system and blood pressure and heart rate are monitored using the finapres. Thereafter, 3.5 hours after the administration of the compound (t=210) BAT activity and volume will be determined using an MRI scan. Furthermore, a venous blood sample will be drawn every 15 minutes to monitor changes in plasma lipids. In addition, plasma catecholamine concentrations will be determined.Study day 3 is exactly the same as study day 2, except this time the subject will receive the other compound (either 200 mg Mirabegron or placebo).

All study days will take place at the Leiden University Medical Centre (LUMC). Between study days 2 and 3 a wash-out period of 13 days will be maintained to make sure that the drug is out of the body during the next exam.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers. 10 white Caucasians, born in the Netherlands. 10 South Asians, living in the Netherlands.
* Age: 18-30 years
* BMI ≤ 25 kg/m2

Exclusion Criteria:

* BMI > 25 kg/m2
* Recent excessive weight loss or exercise
* Alcohol and/ or drugs abuse
* Smoking
* Any significant chronic disease, including diabetes
* Renal, hepatic or endocrine disease
* Heart disease or arrhythmias
* Thyroid disease or thyroid medication
* Hypertension
* Use of medication known to influence glucose and/or lipid metabolism or BAT activity (e.g. beta blockers or calcium channel blockers)
* Use of drugs that influence cardiac function or affect QT time
* Use of MAO inhibitor
* Use of systemic corticosteroids in previous six weeks
* Recent participation in other research projects (within the last 3 months), participation in 2 or more projects in one year
* Contraindications for undergoing an MRI scan:
* Presence of non-MR safe metal implants or objects in the body.
* Pacemaker, neurostimulator, hydrocephalus pump, drug pump, non-removable hearing aid, large recent tattoos.
* Claustrophobia
* Tinnitus or hyperacusis

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The effect of Mirabegron treatment on BAT activity measured by MRI in South Asians compared with white Caucasians. | Up to 1 year
  Brown adipose tissue activity will be measured by means of MRI

SECONDARY OUTCOMES:
Effect of Mirabegron treatment on REE between South Asian and white Caucasian individuals. | Up to 1 year
  Indirect calorimetry will be performed to asses resting energy expenditure
Mild cold exposure and Mirabegron on plasma lipoprotein profiles | Up to 1 year
  Use NMR to analyse lipoproteins in venous blood samples taken during the cooling protocol
Mirabegron treatment on plasma lipid levels between South Asian and white Caucasian individuals. | Up to 1 year
  Use enzymatic assays to determine lipid levels in plasma
The effect of Mirabegron treatment on sympathetic output in South Asian and white Caucasian individuals. | Up to 1 year
  Measure noradrenalin and adrenaline levels in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Jazet, MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

REFERENCES:
- [Derived] Hoekx CA, Martinez-Tellez B, Straat ME, Bizino MB, van Eyk HJ, Lamb HJ, Smit JWA, Jazet IM, Nahon KJ, Janssen LGM, Rensen PCN, Boon MR. Circulating FGF21 is lower in South Asians compared with Europids with type 2 diabetes mellitus. Endocr Connect. 2025 Jan 6;14(2):e240362. doi: 10.1530/EC-24-0362. Print 2025 Feb 1. PMID 39641307
- [Derived] Straat ME, Jurado-Fasoli L, Ying Z, Nahon KJ, Janssen LGM, Boon MR, Grabner GF, Kooijman S, Zimmermann R, Giera M, Rensen PCN, Martinez-Tellez B. Cold exposure induces dynamic changes in circulating triacylglycerol species, which is dependent on intracellular lipolysis: A randomized cross-over trial. EBioMedicine. 2022 Dec;86:104349. doi: 10.1016/j.ebiom.2022.104349. Epub 2022 Nov 11. PMID 36371986